CLINICAL TRIAL: NCT04304560
Title: Value of SGLT2 Inhibitor (Dapagliflozin) as an Added Therapy in Diabetic Patients With Heart Failure With Reduced Ejection Fraction; Randomized Controlled Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Damanhour University (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDHFrEF
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Diabete Type 2; Cardiomyopathies
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiomyopathies | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Control group will receive the standard therapy for DM & HFrEF and placebo.
  Interventions: Drug: Placebo oral tablet
- Dapagliflozin (Experimental): Intervention group will receive 10mg of Dapagliflozin (Forxiga) ® tablet and standard therapy for HFrEF.
  Interventions: Drug: Dapagliflozin 10 MG

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — inhibitor of sodium-glucose cotransporter 2
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo oral tablet — Similar Placebo oral tablet
  Arms: Control Group

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a well-recognized independent risk factor for heart failure (HF). Whereas the prevalence of HF in the general population is 1-4%, it reaches approximately 12% in T2DM patients. In 1972, Rubler reported a specific diabetes-associated cardiac injury called diabetic cardiomyopathy. This cardiomyopathy is defined by ventricular dysfunction occurring without coronary disease or hypertension. Diabetic cardiomyopathy is also characterized by left ventricular (LV) hypertrophy, diastolic dysfunction and myocardial fibrosis.

A large body of work indicates that diabetic cardiomyopathy is associated with altered cardiac energy metabolism. Indeed, in obese T2DM patients, heart lipid uptake is increased. Several studies support that free fatty acid (FFA) accumulation leads to the increased production of diacylglycerol (DAG), ceramides and reactive oxygen species (ROS), affecting cardiac insulin sensitivity and cardiac contractility. On the other hand, hyperglycemia and glucose overload have been involved in cardiac hypertrophy and dysfunction in the context of T2DM and obesity. The diabetic heart is simultaneously characterized by impaired insulin-stimulated glucose uptake and obvious signs of glucose overload, such as ROS and advanced glycation end-product (AGE) production as well as hexosamine pathway chronic activation. Interestingly, when comparing diabetic and nondiabetic obese patients, we previously demonstrated that hyperglycemia per se plays a central role in the impaired cardiac mitochondrial activity associated with myocardial contractile dysfunction.

DETAILED DESCRIPTION:
Primary Objective: The purpose of this study was to investigate the effect of Dapagliflozin, an inhibitor of sodium-glucose cotransporter 2, on cardiovascular Cardiomyopathy, morbidity and mortality in patients with type 2 diabetes.

Secondary Objective: Change in the fibrosis and oxidative stress markers and its relation with progression of cardiomyopathy.

Proposal Steps

1. Ethical committee approval will be obtained from Ethics committee of Faculty of Medicine, Elmenoufia University.
2. This study will be registered at ClinicalTrials.gov after ethical committee approval .
3. All participants should agree to take part in this clinical study and will provide informed consent.
4. 60 participants who are Type 2 Diabetes and HFrEF Patients will be recruited from the Elmenoufia Hospital, Cardiology department, Elmenoufia University,
5. The 60 participants will be randomly assigned into 2 groups:

   * Control groups: receives the standard therapy for DM &HFrEF.
   * The second group: receive 10mg tabs of Dapagliflozin ( Forxiga) ® and standard therapy for HFrEF.
   * Subjects will be treated with medication regimens for at least 3 months
6. All patients will be submitted to:

   * Full patient history and clinical examination.
   * Routine follow up before and after each visit. (complete blood picture, liver function tests, renal function tests).
   * Echocardiography before the start and after completion of the study which include:
   * Conventional echocardiography.
   * All Study participants underwent standard echocardiography with Doppler studies, using a GE vivid 9 machine all subjects were examined in the left lateral Decubitus position according to the recommendations of the American Society of Echocardiography (24).
   * 1) Assessment of LV dimensions:
   * M-mode measurements were obtained from left parasternal with special Attention was given not to include overlying trabeculations in the ventricular septum or posterior wall measurements, which may overestimate thickness.
   * Measurements were taken at the end diastole -defined as the beginning of the QRS complex -but preferably using the widest LV cavity diameter, and at the end systole -using the narrowest LV cavity diameter.
   * The diastolic measurements obtained were the interventricular septal wall thickness, the LV internal diameter at end diastole and posterior wall thickness. In systole, the LV systolic diameter was measured.
   * 2-Systolic function assessment:
   * The measurement of LV ejection fraction (%) and LV fractional shortening (%) were performed to evaluate the systolic function using M mode tracing. Ejection fraction (EF %) was calculated as percentage change of LV chamber volumes between diastole and systole from apical four and two chamber views using modified biplane Simpson's rule. (25)
   * NB: Ejection fraction ≥ 55 % indicated a normal systolic function and <55 % is considered systolic dysfunction.
   * 3-Diastolic Function assessment:
   * Pulsed - wave Doppler echocardiography was used to evaluate diastolic LV function; Doppler studies were recorded from the apical 4- chamber view, with a sample volume positioned with in the inflow portion of the LV, midway between the annular margins of mitral valve. Mitral velocity profiles were digitized from velocity of the Doppler tracings.
   * Waves measured by pulsed conventional Doppler:
   * The peak E (early rapid ventricular filling) wave velocity: It is an early filling wave occurs in the early diastole as the pressure in the left ventricle falls below that in the left atrium (N = 50 - 85 cm / sec).
   * The Peak A (late ventricular filling) wave velocity: It is a late filling wave occurs as the left atrial contraction causes acceleration of the flow from the left atrium to the left ventricle (N = 35 - 5 0 cm/sec). (26)
   * E / A ratio: The ratio between the early filling and the late filling wave (N = 1 - 2).
   * N.B Diastolic dysfunction is considered if DT > 220 ms and E / A ratio < 1.
   * Tissue Doppler Imaging:
   * By using GE Vivid 9 echocardiography machine programmed with tissue Doppler options, tissue Doppler imaging was performed in the apical views (4- chamber, and long axis), continuous wave Doppler tissue imagining was obtained by positioning a sample volume at the basal septal and lateral mitral annuli. Myocardial velocity was detected throughout each cardiac cycle and the average value was recorde
   * Three major velocities were recorded at the annular sites:
   * The peak major positive systolic velocity when the annulus moved towards the apex (Sm) (N = 9.1 ± 1.2 cm/sec).
   * Two peaks of major negative velocities when the annulus moved back towards the base during early (Em) (N = 14.7 ± 314 cm/sec) and late (Am) phase of diastole (N = 11.0 s ± 2.3 cm/sec).
   * E/Em ratio was also calculated.
   * Isovolumic relaxation time (IVRT) is measured from the end of the systolic velocity to the beginning of the early diastolic velocity (N = 59 ± 22 cm/sec).

Systolic dysfunction if peak systolic velocity < 8 cm / sec.

* Diastolic dysfunction is considered if IVRT > 90 ms or E/A<1 or E/Em>10.
* Two-dimensional speckle tracking imaging analysis:
* Parasternal basal and apical short-axis views, as well as three standard apical views, were acquired. All grey scale images were obtained at a frame rate of 77 ± 6 frame/s (range: 63-99 frames/s) using second harmonic imaging. While acquiring images, the LV basal short-axis view was identified by the presence of mitral leaflets, while excluding the mitral annulus and the apical view was identified by the presence of a LV cavity in the absence of papillary muscles. We made every effort to obtain the LV cross-section as circular as possible. For each view, three consecutive cardiac cycles were acquired during a breath hold and digitally stored on a magneto-optical disc for offline analysis. Measurement of strain and rotational parameters was performed offline using dedicated software (Echo-Pac PC, version 10.0; GE Medical systems)
* A region of interest was manually adjusted to include the entire myocardial thickness; care was taken to avoid including the pericardium in the region of interest. The software then selected stable speckles within the myocardium and tracked these speckles frame-by-frame throughout the cardiac cycle. Counterclockwise rotation was marked as a positive value and clockwise rotation as a negative value when viewed from the LV apex. LV twist was defined as the net difference (in degrees) of apical and basal rotations at isochronal time points and was auto computed by the software from the values of the basal and apical rotation. LV torsion was then calculated as the ratio between LV twist (in degrees) and the LV diastolic longitudinal length (in cm) between the LV apex and the mitral plane.
* A pulse wave Doppler tracing obtained from the LV outflow tract was used to identify the timing of aortic valve opening and closure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with type-2 diabetes history >=5 years
2. HbA1C 6-10% with glucose control medications including insulin, metformin or sulfonylurea
3. Medically stable
4. Willing to participate and sign informed consent.

Exclusion Criteria:

1. GFR <60 mL/min/1.73 m2
2. Unstable or rapidly progressive renal disease
3. Hypotension with SBP <100 mmHg
4. Hypersensitivity to dapagliflozin or any excipients
5. Patients with severe hepatic impairment (Child-Pugh class C)
6. Patients with active hepatitis B or C infection
7. Any of the following CV/Vascular Diseases within 3 months prior to signing the consent at enrollment, as assessed by the investigator:

   1. Myocardial infarction
   2. Cardiac surgery or revascularization (CABG/PTCA)
   3. Unstable angina
   4. HF New York Heart Association (NYHA) Class IV
   5. Transient ischemic attack (TIA) or significant cerebrovascular disease
   6. Unstable or previously undiagnosed arrhythmia
   7. Established PAD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
LV dimensions | 3 Months
  Echocardiography
Systolic function | 3 Months
  Echocardiography
Diastolic Function | 3 Months
  Echocardiography

SECONDARY OUTCOMES:
HbA1c | 3 Months
  Glycemic control
Myeloperoxidase (MPO) | 3 Months
  Oxidative stress marker
N-terminal pro b-type Natriuretic Peptide (proBNP-N) | 3 Months
  Fibrosis marker
Galectin -3 | 3 Months
  Fibrosis marker

IPD SHARING:
Plan to Share IPD: Undecided